CLINICAL TRIAL: NCT05292482
Title: Pragmatic Randomized Controlled Trial of Pharmacopuncture Therapy for Adhesive Capsulitis : A Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jaseng Hospital of Korean Medicine (Other)
Collaborators: Korea Institute of Oriental Medicine (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: JS-CT-2022-01
Record Dates: First submitted 2022-03-15; First posted 2022-03-23 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2022-12

CONDITIONS: Adhesive Capsulitis
MeSH Terms: conditions — Bursitis | interventions — Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- pharmacopunture therapy (Experimental): The physicians will choose the type and volume of pharmacopuncture according to participants' conditions and inject it at the proper acupoints they choose.
  Interventions: Procedure: pharmacopuncture therapy
- physical therapy (Active Comparator): The physicians will choose the type and time of physical therapy according to participants' conditions.
  Interventions: Procedure: physical therapy

INTERVENTIONS:
Procedure: pharmacopuncture therapy — This is a pragmatic RCT, so the physicians will choose the type and volume of pharmacopuncture according to participants' conditions.
  Arms: pharmacopunture therapy
Procedure: physical therapy — This is a pragmatic RCT, so the physicians will choose the type and time of physical therapy according to participants' conditions.
  Arms: physical therapy

SUMMARY:
This is a 2-arm parallel pragmatic randomized controlled trial that will compare pharmacopuncture therapy with physical therapy for adhesive capsulitis.

DETAILED DESCRIPTION:
Participants who voluntarily signed informed consent form and eligible for the study were randomly assigned in a 1:1 ratio (25:25) for pharmacopuncture therapy and physical therapy group. Participants of each group will receive twice a week for total 6 weeks of intervention. This is a pragmatic randomized controlled trial, so physicians will have medical decision making according to each participant's conditions.

ELIGIBILITY:
Inclusion Criteria:

* Limitation of the shoulder movement (active or passive)
* Numeric Rating Scale (NRS) of neck pain is more than 5
* Symptoms of adhesive capsulitis for more than 1 month
* Discrimination findings which can explain clinical symptoms on shoulder MRI or CT
* 19-69 years old
* participants who agreed and wrote informed consents

Exclusion Criteria:

* Case of being diagnosed with a specific serious disease that may cause shoulder pain(Fracture, Dislocation, etc.)
* Cause of pain due to soft tissue disease, not the spine(Cancer, fibromyalgia, RA, goat, or etc.) Other chronic diseases(stroke, MI, kidney disease, diabetic neuropathy, dimentia, epilepsy, or etc.) that may interfere with the interpretation of therapeutic effects or outcomes
* Participants taking steroid, immunosuppressant, psychotropic medication, or taking other drugs that may affect outcomes
* Inappropriate or unsafe pharmacopuncture therapy; hemorrhagic disease, taking anticoagulant drug, or severe diabetes patients who are likely to be infected
* Participants who took NSAIDs or pharmacopuncture, acupuncture, physical therapy within 1 week
* Pregnant, planning to get pregnant or lactating women
* Participants who had undergone shoulder surgery within 3 months
* Participants who had participated in other clinical trial within 1 month, had participated in other study within 6 months from the date of selection, or have plan for participation in other trial during follow up period of this trial
* Participants who can not write informed consent
* Participants who is difficult to participate in the trial according to investigator's decision

Ages: 19 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2022-04-20 (Actual); Primary Completion 2022-10-25 (Actual); Study Completion 2022-12-06 (Actual)

PRIMARY OUTCOMES:
Numeric rating scale (NRS) of shoulder pain | week 7
  NRS is a pain scale in which the patient indicates their subjective pain as a whole number from 0 to 10, where 0 indicates 'no pain or discomfort' and 10 indicates 'the most severe pain and discomfort imaginable'.

SECONDARY OUTCOMES:
Visual analogue scale (VAS) of shoulder pain | week 1, 2, 3, 4, 5, 6, 7, 13
  Visual analogue scale of shoulder pain, minimum 0 to maximum 100, which is a higher score means a worse outcome.
ROM(Range of motion) | week 1, 2, 3, 4, 5, 6, 7, 13
  The range of shoulder movement shows the function of the shoulder capsule.
SPADI | week 1, 7, 13
  SPADI is a functional disability questionnaire. The possible range of each item score is 0 to 10. Total score range is 0 (better outcome) to 100 (worse outcome).
PGIC | week 7, 13
  Participants rate the improvement after treatment on a 7-point Likert scale (1, very much improved; 2, much improved; 3, minimally improved; 4, no change; 5, minimally worse; 6, much worse; or 7, very much worse.)
SF-12 v2 | week 1, 7, 13
  The SF-12 consists of 12 questions across 8 domains, and higher scores indicate better health-related quality of life.
EQ-5D-5L | week 1, 7, 13
  The EQ-5D-5L consists of 5 questions (mobility, self-care, usual activities, pain, anxiety/depression) that ask about the current state of health, and answers each question with 5 likert. (1=I have no problems about, 2=I have slight problems about, 3=I have moderate problems about, 4=I have severe problems about, 5=I am unable to about)

CONTACTS AND LOCATIONS:
Overall Officials: Kyoung Sun Park, Ph.D, Principal Investigator — Jaseng Hospital of Korean Medicine
Locations (1):
- Jaseng Korean Medicine Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kim D, Park KS, Kim SA, Seo JY, Cho HW, Lee YJ, Yang C, Ha IH, Han CH. Pharmacopuncture therapy for adhesive capsulitis: A pragmatic randomized controlled pilot study. Integr Med Res. 2024 Sep;13(3):101065. doi: 10.1016/j.imr.2024.101065. Epub 2024 Jun 21. PMID 39224580